CLINICAL TRIAL: NCT05341882
Title: Adaptation of Mindfulness Training to Treat Moral Injury in Veterans
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Old Dominion University (Other)
Collaborators: William & Mary (Other); H. Lee Moffitt Cancer Center and Research Institute (Other); University of North Carolina, Chapel Hill (Other)
Responsible Party: Principal Investigator, Michelle L. Kelley, Professor of Psychology, Old Dominion University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0414484650000
Record Dates: First submitted 2021-09-14; First posted 2022-04-22 (Actual); Last update posted 2023-06-05 (Actual); Status verified 2023-05

CONDITIONS: Mindfulness; Educational Support
Keywords: Mindfulness; Veterans; Moral Injury; Educational Support
MeSH Terms: conditions — Stress Disorders, Post-Traumatic | interventions — Mindfulness; Training Support

STUDY DESIGN:
Intervention Model Description: In Study 2, we randomized 19 participants to either the Mindfulness or Educational Support condition. In Study 3, we randomized 56 participants to the Mindfulness or Educational Support condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mindfulness (Experimental): The seven weekly sessions teach veterans how to use mindfulness techniques in everyday life and when dealing with stress and negative emotions related to moral injury.
  Interventions: Behavioral: Mindfulness
- Educational Support (Active Comparator): As an active control condition, the investigators developed an education support (ES) group, which ran concurrently to the mindfulness intervention group. Within the military community, peer support and psychoeducation are considered critical components of alleviation of suffering from traumatic exposure.
  Interventions: Behavioral: Educational Support

INTERVENTIONS:
Behavioral: Mindfulness — Participants took part in a live, facilitated Zoom-delivered training that involved learning mindfulness and education about moral injury. The participants were interviewed regarding the program.
  Arms: Mindfulness
Behavioral: Educational Support — As an active control condition, the investigators developed an education support (ES) group, which ran concurrently to the mindfulness intervention group. Within the military community, peer support and psychoeducation are considered critical components of alleviation of suffering from traumatic exposure.
  Arms: Educational Support

SUMMARY:
This project is highly innovative as it will be the first to develop a mindfulness-based treatment as a first-line intervention tailored to target moral injury among combat-wounded veterans. In Study 1, the investigators recruited a small group of veterans to give feedback on the project. In Studies 2 and 3, the investigators will compare the newly developed mindfulness training to an equally intensive Educational Support condition. Further, if successful, this application may have the ability to adapted and extended to address common to other professions that experience moral injury.

DETAILED DESCRIPTION:
Combat theaters place service members in situations where they make difficult decisions that may transgress deeply held moral beliefs or witness others' acts of betrayal. Although many veterans are resilient to these types of experiences, for others, failure to accommodate these events may result in internal conflict that is theorized to lead to the development of moral injury. Moral injury is distinct from posttraumatic stress disorder and has been associated with poor mental health outcomes (e.g., depression, anxiety, suicidality) and alcohol/drug use among veterans. Few evidence-based interventions have been developed to target symptoms of moral injury. In studies with combat wounded veterans, community veterans, and a predominantly VA treatment-seeking sample, the investigators have demonstrated that mindfulness moderates associations between moral injury symptoms and negative mental health outcomes. In addition, the investigators have demonstrated that combat wounded veterans are willing to take part in a mindfulness-based moral injury intervention, especially if administered in an online interactive web-based program. Using an iterative developmental process, the goal of this project is to adapt an integrative and theory-driven mindfulness-based intervention delivered online to target moral injury in combat wounded veterans. Aim 1 is to modify an evidence-based, online, interactive, instructor-delivered, six-session mindfulness program, originally designed to help active duty members manage physical pain (i.e., Mindfulness to Manage Chronic Pain), such that it addresses the psychologically painful symptoms (e.g., guilt, shame) characteristic of those with moral injury. The newly adapted program, Mindfulness to Manage Moral Injury (MMMI), will then be piloted with one group of eligible veterans (N = 6) to generate qualitative feedback on program content and format; revisions based on this feedback will result in preliminary manualization. Subsequently, in Aim 2 the investigators propose to develop a facilitator-led online interactive Education Support (ES) program designed to serve as a control comparison intervention, and then carry out a non-randomized pilot study comparing the feasibility (i.e., credibility, acceptability, study completion, and adherence (e.g., to homework assignments) of ES to the revised MMMI program with N = 20 (10 MMMI; 10 ES) recent-era veterans. Following this phase of feasibility testing, the investigative team will collect qualitative information and further refine both the MMMI and ES materials. In Aim 3, the investigators propose a small-scale randomized controlled trial (N = 42 combat wounded veterans; 21 MMMI; 21 ES) to collect data on recruitment, credibility and acceptability, completion rates, and adherence in the two newly refined intervention arms at pre-post-test. Aim 3 will assess for potential primary and secondary outcome measures and lay the groundwork for a large-scale randomized R01 controlled efficacy trial. If supported, this work would have the potential to provide a novel and flexible theoretically grounded form of treatment delivered in-home for combat wounded veterans experiencing moral injury symptoms and associated mental health problems.

ELIGIBILITY:
Inclusion Criteria:

1. Post 9/11 veterans who were deployed to Iraq/Afghanistan regions 1 or more times
2. Report 2 or more symptoms of moral injury

Exclusion Criteria:

1. They have a probable psychotic disorder (as determined by the Diagnostic and Statistical Manual-5 Level 1 Cross-Cutting Symptom Measure-Adult)

   or
2. They have a current suicide plan

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as male or female.
Enrollment: 75 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2022-10-19 (Actual); Study Completion 2022-10-19 (Actual)

PRIMARY OUTCOMES:
Semi-Structured Interviews | 1 hour
  Semi-structured interview to obtain input on the study programs

CONTACTS AND LOCATIONS:
Overall Officials: Michelle L Kelley, Ph.D., Principal Investigator — Old Dominion University
Locations (1):
- Old Dominion University, Norfolk, Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Given this is an R34 grant, we developed a mindfulness program via an iterative process. We then completed a protocol paper that describes the development process and the mindfulness and active control training programs.

REFERENCES:
- [Background] Kelley ML, Strowger M, Chentsova VO, Bravo AJ, Gaylord SA, Burgin EE, Vinci C, Ayers KL, Agha E. Mindfulness to Manage Moral Injury: Rationale and development of a live online 7-week group intervention for veterans with moral injury. Contemp Clin Trials Commun. 2022 Oct 14;30:101011. doi: 10.1016/j.conctc.2022.101011. eCollection 2022 Dec. PMID 36340697

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/82/NCT05341882/Prot_SAP_000.pdf